CLINICAL TRIAL: NCT01749865
Title: A Randomized Controlled Study of Cytokine-induced Killer Cell (CIK) Treatment in Patients With Hepatocellular Carcinoma Who Underwent Radical Resection
Brief Title: CIK Treatment for HCC Patient Underwent Radical Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, LI Sheng-ping, Vice director, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007043-HCC012
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A, CIK (Experimental): Biological/Vaccine: Cytokine-Induced Killer Cells
  Interventions: Biological: Cytokine-Induced Killer Cells
- B, CONTROL (No Intervention): Regular follow up with no intervention

INTERVENTIONS:
Biological: Cytokine-Induced Killer Cells — Cytokine-Induced Killer Cells treatment for 4 cycles
  Other Names: CIK
  Arms: A, CIK

SUMMARY:
This is a randomized controlled study. About 200 patients with hepatocellular carcinoma who underwent radical resection will be included. The patients will be randomized to group A (receive CIK treatment) or group B (just regularly follow up) without any anti-cancer treatment after resection of HCC, and the randomize ratio will be 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age.
* Without any prior anti-cancer therapy.
* Patients who have a life expectancy of at least 12 weeks.
* Patients already had radical resection of HCC.

Definition of radical resection in this study:

* All tumors were moved out, with a clean resection margin.
* Number of tumors less than 3.
* Without tumor invasion of the main trunk and first branch of the portal vein, or hepatic duct, or hepatic vein.
* No hepatic hilum lymphnode metastasis.
* No distance metastasis.
* Hepatocellular carcinoma with histological diagnose.
* No major post-operative complication.
* Patients who have an performance status of 0, or 1.
* Cirrhotic status of Child-Pugh class A only.
* The following laboratory parameters:
* Patients who give written informed consent.

Exclusion Criteria:

* Previous or concurrent cancer that is distinct in primary site or histology from HCC.
* History of cardiac disease.
* Active clinically serious infections ( over grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* History of organ allograft.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial.
* Pregnant or breast-feeding patients.
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study.
* Excluded therapies and medications, previous and concomitant:

Prior use of any anti-cancer treatment for HCC, eg. chemotherapy, radiotherapy. Antiviral treatment is allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | 5-year
  To evaluate efficacy of CIK treatment as an adjuvant therapy in patients with hepatocellular carcinoma (HCC) who underwent radical resection.

SECONDARY OUTCOMES:
Disease Free Survival | 5 year
  Disease Free Survival

OTHER OUTCOMES:
Adverse Events | 5 years
  To evaluate safety of CIK treatment as an adjuvant therapy in patients with hepatocellular carcinoma (HCC) who underwent radical resection.

CONTACTS AND LOCATIONS:
Locations (1):
- Immunotherapy, Guangzhou, Guangdong, China